CLINICAL TRIAL: NCT00478608
Title: A Clinical Study to Evaluate the Efficacy and Safety of Cyclosporine (CsA) and Sirolimus (SRL) Induction Followed by Cyclosporine Withdrawal in Korean Renal Allograft Recipients
Brief Title: Study Evaluating Rapamune® Maintenance Regimen
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Wyeth (Registry Contact: Clinical Trial Registry Specialist), Wyeth
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 0468E-102362
Record Dates: First submitted 2007-05-24; First posted 2007-05-25 (Estimated); Results first posted 2010-01-07 (Estimated); Last update posted 2010-04-28 (Estimated); Status verified 2010-04

CONDITIONS: Renal Transplant
MeSH Terms: interventions — Sirolimus

INTERVENTIONS:
Drug: Sirolimus (Rapamune®) — (1mg tablets): Initial loading dose of 6mg/day, followed by maintenance dose of 2mg/day, which was adjusted to specified trough level.

SUMMARY:
Primary : To evaluate the efficacy of sirolimus assessed by the incidence of biopsy-confirmed acute rejection episode at 6 months after transplantation in Korean renal transplantation recipients.

Secondary :

1. To evaluate the safety of sirolimus over 12 months after transplantation in Korean renal transplantation recipients.
2. To evaluate graft function, patient survival and graft survival at 6 and 12 months after transplantation, and to investigate the incidence of biopsy-confirmed acute rejection episode at 12 months after transplantation.

ELIGIBILITY:
Inclusion Criteria:

1. Age greater than or equal to 13 years of age.
2. End-stage renal disease in patients scheduled to receive a primary renal allograft from a cadaveric donor, a living-unrelated donor, or from a living-related (excluding 0 antigen mismatch) donor. A mismatch donor is defined as a donor human leukocyte antigen (HLA) antigen not shared by the patient.
3. Patients with a panel of reactive antibody (%PRA) less than or equal to 50%

Exclusion Criteria:

1. Evidence of active systemic or localized major infection at the time of initial sirolimus administration.
2. Evidence of infiltrate, cavitation, or consolidation on chest x-ray obtained during pre-study screening.
3. Chronic anti-arrhythmic therapy for ventricular arrhythmia or other cardiac abnormality contraindicating general anesthesia or surgery.
4. History of malignancy within 5 years before enrollment into the study (with the exception of adequately treated basal cell or squamous cell carcinoma of the skin).
5. Current treatment with partial opioid agonists (eg, buprenorphine) or combination agonists/antagonists.

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2007-03; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer
Locations (4):
- South Korea (4):
  - Deagu
  - Pusan
  - Seoul
  - Suwon

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited in Korea from March 2007 to November 2007.
Pre-assignment Details: Patients were screened up to 7 days.
Groups:
- Sirolimus (SRL): Patients initially received SRL, Cyclosporine (CsA) and Corticosteroids. After 2-4 months following transplantation, CsA was progressively withdrawn.
  On Day 1 (within 48 hours after transplantation) SRL was initiated (6 mg loading dose). For Day 2 through CsA withdrawal (w/d), SRL dose was 2mg/day, with adjustment to maintain a target trough blood level of 5-15 ng/ml. During CsA w/d through month 6, SRL dose adjusted to a trough level of 15-30 ng/ml; and for months 7-12, a trough level of 12-24 ng/ml.
  CsA initiated before or within 48 hours after transplantation at a dose to attain a trough level of 200-400 ng/ml. From month 1 to time of CsA w/d, CsA dose was adjusted to maintain a trough level of 150-300 ng/ml. At 2 to 4 months after transplantation, CsA was withdrawn over 4-8 weeks.
  Corticosteroids were initiated within 24 hours before or after transplantation and tapered to ≥ 5 mg/day of prednisone by the end of week 13. W/d of corticosteroids was prohibited.
Period: Overall Study
Arm/Group | Sirolimus (SRL)
Started | 79
Completed | 59
Not Completed | 20
Not completed — Adverse Event | 1
Not completed — Serious Adverse Event | 14
Not completed — Withdrawal by Subject | 2
Not completed — Protocol Violation | 3

BASELINE CHARACTERISTICS:
Arm/Group | Sirolimus (SRL)
Number analyzed (Participants) | 79
Age Continuous [Mean (Standard Deviation); unit: years] | 40.16 (12.69)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 47
  Male | 32

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients Experiencing Biopsy Confirmed Acute Rejection Through Month 6 After Transplantation.
Description: The diagnosis of acute rejection required a kidney biopsy. Biopsies were assessed using the Banff criteria, standardized diagnostic categories based on histological assessments (e.g., cell types and distributions).
Time Frame: 6 months after transplantation
Population: Patients who received at least one dosing of SRL after transplantation.
Measure: Number; unit: patients
Arm/Group | Sirolimus (SRL)
Number analyzed (Participants) | 79
patients | 12

2. Secondary Outcome: Glomerular Filtration Rate (GFR) (Nankivell Method)
Description: GFR is an index of kidney function. GFR describes the flow rate of filtered fluid through the kidney. GFR can be measured directly or estimated using established formulas. For this study, GFR was calculated using the Nankivell formula. A normal GFR is >90 mL/min, although children and older people usually have a lower GFR. Lower values indicate poorer kidney function. A GFR <15 is consistent with kidney failure.
Time Frame: 6 and 12 months
Population: Patients who received at least one dose of SRL after transplantation. Observed values
Measure: Mean (Standard Deviation); unit: mL/min
Arm/Group | Sirolimus (SRL)
Number analyzed (Participants) | 79
mL/min
  6 months | 67.36 (15.25)
  12 months | 71.92 (18.82)

3. Secondary Outcome: Serum Creatinine
Description: Serum creatinine is an indicator of kidney function. Creatinine is a substance formed from the metabolism of creatine, commonly found in blood, urine, and muscle tissue. It is removed from the blood by the kidneys and excreted in urine. An increased level of creatinine in the blood indicates decreased kidney function. Normal adult blood levels of creatinine are 0.5 to 1.1 mg/dL for females and 0.6 to 1.2 mg/dL for males; however, the normal values are age-dependent as elderly patients typically have smaller muscle mass.
Time Frame: Baseline, 6 and 12 months
Population: Patients who received at least one dose of SRL after transplantation. Observed values
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Sirolimus (SRL)
Number analyzed (Participants) | 79
mg/dl
  Baseline | 9.42 (3.64)
  6 months | 1.30 (0.36)
  12 months | 1.25 (0.43)

4. Secondary Outcome: Patient and Graft Survival
Description: Patient survival defined as patients living with or without a functioning graft. Graft survival defined as those patients who did not experience graft loss. Graft loss defined as physical loss (nephrectomy), functional loss (necessitating maintenance dialysis for >8 weeks), retransplant or death during the first 12 months after randomization.
Time Frame: 12 months
Population: Patients who received at least one dosing of SRL after transplantation.
Measure: Number; unit: patients
Arm/Group | Sirolimus (SRL)
Number analyzed (Participants) | 79
patients
  Patient survival 6 months | 77
  Patient survival 12 months | 76
  Graft survival 6 months | 77
  Graft survival 12 months | 76

5. Secondary Outcome: Number of Patients Experiencing Biopsy Confirmed Acute Rejection Through Month 12 After Transplantation
Description: as for outcome 1
Time Frame: 12 months after transplantation
Population: Patients who received at least one dosing of SRL after transplantation.
Measure: Number; unit: patients
Arm/Group | Sirolimus (SRL)
Number analyzed (Participants) | 79
patients | 15

ADVERSE EVENTS:
Arm/Group | Sirolimus (SRL)
Serious Adverse Events (participants affected / at risk) | 39/79
Other Adverse Events (participants affected / at risk) | 79/79
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sirolimus (SRL) (N=79)
Herpes zoster (Infections and infestations) | 6
Pneumonia (Infections and infestations) | 5
Gastroenteritis (Infections and infestations) | 2
Urinary tract infection (Infections and infestations) | 2
Varicella (Infections and infestations) | 1
Parotitis (Infections and infestations) | 1
Pulmonary tuberculosis (Infections and infestations) | 1
Enterocolitis infectious (Infections and infestations) | 1
Fungal infection (Infections and infestations) | 1
Cellulitis (Infections and infestations) | 1
Blood creatinine increased (Investigations) | 10
Aspartate aminotransferase increased (Investigations) | 1
Blood glucose increased (Investigations) | 1
Alanine aminotransferase increased (Investigations) | 1
Diarrhoea (Gastrointestinal disorders) | 3
Abdominal pain (Gastrointestinal disorders) | 1
Abdominal hernia (Gastrointestinal disorders) | 1
Inguinal hernia (Gastrointestinal disorders) | 1
Haematochezia (Gastrointestinal disorders) | 1
Faecaloma (Gastrointestinal disorders) | 1
Lymphocele (Vascular disorders) | 6
Pyrexia (General disorders) | 2
Oedema peripheral (General disorders) | 1
Oedema (General disorders) | 1
Asthenia (General disorders) | 1
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1
Asphyxia (Respiratory, thoracic and mediastinal disorders) | 1
Myocardial infarction (Cardiac disorders) | 1
Cardiac failure congestive (Cardiac disorders) | 1
Myocarditis (Cardiac disorders) | 1
Haemolytic uraemic syndrome (Blood and lymphatic system disorders) | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 2
Urinary incontinence (Renal and urinary disorders) | 1
Renal mass (Renal and urinary disorders) | 1
Seroma (Injury, poisoning and procedural complications) | 1
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1
Cervix carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Death (General disorders) | 3
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sirolimus (SRL) (N=79)
Constipation (Gastrointestinal disorders) | 31
Diarrhoea (Gastrointestinal disorders) | 21
Nausea (Gastrointestinal disorders) | 16
Mouth ulceration (Gastrointestinal disorders) | 14
Vomiting (Gastrointestinal disorders) | 13
Abdominal pain (Gastrointestinal disorders) | 12
Dyspepsia (Gastrointestinal disorders) | 8
Abdominal pain upper (Gastrointestinal disorders) | 7
Abdominal discomfort (Gastrointestinal disorders) | 5
Stomatitis (Gastrointestinal disorders) | 5
Abdominal distension (Gastrointestinal disorders) | 4
Gingival hyperplasia (Gastrointestinal disorders) | 2
Epigastric discomfort (Gastrointestinal disorders) | 1
Haematemesis (Gastrointestinal disorders) | 1
Oral disorder (Gastrointestinal disorders) | 1
Gastrointestinal disorder (Gastrointestinal disorders) | 1
Oral discomfort (Gastrointestinal disorders) | 1
Faecal incontinence (Gastrointestinal disorders) | 1
Dental caries (Gastrointestinal disorders) | 1
Anorectal disorder (Gastrointestinal disorders) | 1
Abdominal pain lower (Gastrointestinal disorders) | 1
Blood cholesterol increased (Investigations) | 29
Alanine aminotransferase increased (Investigations) | 17
Aspartate aminotransferase increased (Investigations) | 12
Urine output decreased (Investigations) | 11
Blood lactate dehydrogenase increased (Investigations) | 10
Blood creatinine increased (Investigations) | 9
Hepatic enzyme increased (Investigations) | 9
Blood triglycerides increased (Investigations) | 8
Blood glucose increased (Investigations) | 8
Weight increased (Investigations) | 5
Blood pressure increased (Investigations) | 4
Blood phosphorus decreased (Investigations) | 3
Haemoglobin decreased (Investigations) | 3
Blood albumin decreased (Investigations) | 3
Blood potassium increased (Investigations) | 2
Blood uric acid increased (Investigations) | 2
Body temperature increased (Investigations) | 1
Platelet count decreased (Investigations) | 1
Blood potassium decreased (Investigations) | 1
Gamma-glutamyltransferase increased (Investigations) | 1
Blood calcium decreased (Investigations) | 1
Blood alkaline phosphatase increased (Investigations) | 1
Blood calcium increased (Investigations) | 1
White blood cells urine positive (Investigations) | 1
White blood cell count decreased (Investigations) | 1
Upper respiratory tract infection (Infections and infestations) | 26
Nasopharyngitis (Infections and infestations) | 12
Urinary tract infection (Infections and infestations) | 6
Herpes zoster (Infections and infestations) | 6
Herpes simplex (Infections and infestations) | 4
Rhinitis (Infections and infestations) | 2
Oral candidiasis (Infections and infestations) | 2
Tinea versicolour (Infections and infestations) | 2
Tinea pedis (Infections and infestations) | 2
Varicella (Infections and infestations) | 1
Vaginal infection (Infections and infestations) | 1
Tinea cruris (Infections and infestations) | 1
Folliculitis (Infections and infestations) | 1
Bacteraemia (Infections and infestations) | 1
BK virus infection (Infections and infestations) | 1
Infection (Infections and infestations) | 1
Skin infection (Infections and infestations) | 1
Rash pustular (Infections and infestations) | 1
Gingival infection (Infections and infestations) | 1
Fungal infection (Infections and infestations) | 1
Gastroenteritis (Infections and infestations) | 1
Orchitis (Infections and infestations) | 1
Hypercholesterolaemia (Metabolism and nutrition disorders) | 19
Hyperlipidaemia (Metabolism and nutrition disorders) | 12
Hyperkalaemia (Metabolism and nutrition disorders) | 8
Hypokalaemia (Metabolism and nutrition disorders) | 6
Hypoalbuminaemia (Metabolism and nutrition disorders) | 5
Hyperglycaemia (Metabolism and nutrition disorders) | 5
Diabetes mellitus (Metabolism and nutrition disorders) | 4
Hypophosphataemia (Metabolism and nutrition disorders) | 2
Hyponatraemia (Metabolism and nutrition disorders) | 2
Hypoglycaemia (Metabolism and nutrition disorders) | 2
Hypocalcaemia (Metabolism and nutrition disorders) | 1
Electrolyte imbalance (Metabolism and nutrition disorders) | 1
Anorexia (Metabolism and nutrition disorders) | 1
Hyperamylasaemia (Metabolism and nutrition disorders) | 1
Pyrexia (General disorders) | 8
Chest discomfort (General disorders) | 7
Oedema peripheral (General disorders) | 6
Generalised oedema (General disorders) | 5
Oedema (General disorders) | 5
Pitting oedema (General disorders) | 2
Face oedema (General disorders) | 2
Chest pain (General disorders) | 2
Catheter site pain (General disorders) | 1
Mass (General disorders) | 1
Influenza like illness (General disorders) | 1
Swelling (General disorders) | 1
Sense of oppression (General disorders) | 1
Xerosis (General disorders) | 1
Acne (Skin and subcutaneous tissue disorders) | 18
Pruritus (Skin and subcutaneous tissue disorders) | 10
Rash (Skin and subcutaneous tissue disorders) | 7
Hirsutism (Skin and subcutaneous tissue disorders) | 2
Rash papular (Skin and subcutaneous tissue disorders) | 1
Ecchymosis (Skin and subcutaneous tissue disorders) | 1
Periorbital oedema (Skin and subcutaneous tissue disorders) | 1
Neurodermatitis (Skin and subcutaneous tissue disorders) | 1
Skin disorder (Skin and subcutaneous tissue disorders) | 1
Dry skin (Skin and subcutaneous tissue disorders) | 1
Dermal cyst (Skin and subcutaneous tissue disorders) | 1
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 1
Rash macular (Skin and subcutaneous tissue disorders) | 1
Blister (Skin and subcutaneous tissue disorders) | 1
Alopecia (Skin and subcutaneous tissue disorders) | 1
Toxic skin eruption (Skin and subcutaneous tissue disorders) | 1
Swelling face (Skin and subcutaneous tissue disorders) | 1
Procedural pain (Injury, poisoning and procedural complications) | 24
Post procedural complication (Injury, poisoning and procedural complications) | 2
Postoperative wound complication (Injury, poisoning and procedural complications) | 1
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1
Femur fracture (Injury, poisoning and procedural complications) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 11
Arthralgia (Musculoskeletal and connective tissue disorders) | 6
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 2
Osteoporosis (Musculoskeletal and connective tissue disorders) | 2
Neck pain (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1
Coccydynia (Musculoskeletal and connective tissue disorders) | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 1
Headache (Nervous system disorders) | 15
Convulsion (Nervous system disorders) | 3
Dizziness (Nervous system disorders) | 2
Paraesthesia (Nervous system disorders) | 2
Tremor (Nervous system disorders) | 2
Neuropathy peripheral (Nervous system disorders) | 1
Neuralgia (Nervous system disorders) | 1
Migraine (Nervous system disorders) | 1
Somnolence (Nervous system disorders) | 1
Hypoaesthesia (Nervous system disorders) | 1
Dysarthria (Nervous system disorders) | 1
Anaemia (Blood and lymphatic system disorders) | 19
Leukopenia (Blood and lymphatic system disorders) | 4
Neutropenia (Blood and lymphatic system disorders) | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1
Leukocytosis (Blood and lymphatic system disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 8
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 7
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 6
Productive cough (Respiratory, thoracic and mediastinal disorders) | 3
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 2
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1
Insomnia (Psychiatric disorders) | 12
Sleep disorder (Psychiatric disorders) | 2
Haematuria (Renal and urinary disorders) | 7
Proteinuria (Renal and urinary disorders) | 3
Azotaemia (Renal and urinary disorders) | 2
Albuminuria (Renal and urinary disorders) | 1
Pollakiuria (Renal and urinary disorders) | 1
Renal tubular necrosis (Renal and urinary disorders) | 1
Amenorrhoea (Reproductive system and breast disorders) | 4
Ovarian cyst (Reproductive system and breast disorders) | 2
Erectile dysfunction (Reproductive system and breast disorders) | 2
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1
Vaginal haemorrhage (Reproductive system and breast disorders) | 1
Genital haemorrhage (Reproductive system and breast disorders) | 1
Dysmenorrhoea (Reproductive system and breast disorders) | 1
Visual disturbance (Eye disorders) | 2
Vision blurred (Eye disorders) | 1
Xerophthalmia (Eye disorders) | 1
Ocular hyperaemia (Eye disorders) | 1
Conjunctivitis (Eye disorders) | 1
Dry eye (Eye disorders) | 1
Eyelid oedema (Eye disorders) | 1
Conjunctival oedema (Eye disorders) | 1
Hypertension (Vascular disorders) | 6
Lymphocele (Vascular disorders) | 1
Arrhythmia (Cardiac disorders) | 2
Palpitations (Cardiac disorders) | 1
Myocardial infarction (Cardiac disorders) | 1
Angina pectoris (Cardiac disorders) | 1
Hyperthyroidism (Endocrine disorders) | 2
Cushingoid (Endocrine disorders) | 2
Hepatitis (Hepatobiliary disorders) | 2
Hepatotoxicity (Hepatobiliary disorders) | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 1
Hypoacusis (Ear and labyrinth disorders) | 1
Ear pain (Ear and labyrinth disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PIs agreed to allow the sponsor 60 days to review and require changes to presentations or publications but only to protect confidential information and intellectual property, and for the sponsor to file a patent application, as applicable. The PIs also agreed for data to be presented first as a joint, multi-center publication.